CLINICAL TRIAL: NCT04608630
Title: Bone Loss Prevention With Zoledronic Acid or Denosumab in Critically Ill Adults - A Randomised Controlled Trial
Brief Title: Bone Loss Prevention With Zoledronic Acid or Denosumab in Critically Ill Adults
Acronym: BoneZone
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANZIC-RC/NO001
Record Dates: First submitted 2020-10-25; First posted 2020-10-29 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Critical Illness; Osteoporosis
Keywords: Intensive Care Unit; Osteoporosis; Bone densitometry; Zoledronic acid; Denosumab
MeSH Terms: conditions — Critical Illness; Osteoporosis | interventions — Denosumab; Zoledronic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Denosumab (Active Comparator): Patients allocated to the Denosumab arm will receive Denosumab 60mg in 1ml, administered via subcutaneous injection on Study Days 1 and 180.
  Interventions: Drug: Denosumab 60 MG/ML; Drug: Sodium Chloride 0.9% or 5% Dextrose Intravenous
- Zoledronic acid (Active Comparator): Patients allocated to the Zoledronic acid arm will receive Zoledronic acid 5mg in 100ml 0.9% Sodium Chloride or 5% Dextrose, administered via intravenous infusion over at least 15 minutes on Study Day 1.
  Interventions: Drug: Zoledronic Acid 5Mg/Bag 100Ml Inj; Drug: Sodium Chloride 0.9% Injection
- Placebo (Placebo Comparator): Patients allocated to the placebo arm will receive 0.9% Sodium Chloride 1ml administered via subcutaneous injection on Days 1 and Day 180 and 0.9% Sodium Chloride 100ml or 5% Dextrose administered via intravenous infusion over at least 15 minutes on Day 1.
  Interventions: Drug: Sodium Chloride 0.9% or 5% Dextrose Intravenous; Drug: Sodium Chloride 0.9% Injection

INTERVENTIONS:
Drug: Denosumab 60 MG/ML — Patients allocated to the Denosumab arm will receive Denosumab 60mg in 1ml, administered via subcutaneous injection on Study Days 1 and 180.
  Other Names: Prolia; Xgeva
  Arms: Denosumab
Drug: Zoledronic Acid 5Mg/Bag 100Ml Inj — Patients allocated to the Zoledronic acid arm will receive Zoledronic acid 5mg in 100ml 0.9% Sodium Chloride or 5% Dextrose, administered via intravenous infusion over at least 15 minutes on Study Day 1.
  Other Names: Zometa; Reclast; Aclasta
  Arms: Zoledronic acid
Drug: Sodium Chloride 0.9% or 5% Dextrose Intravenous — Patients allocated to the placebo arm and Denosumab arm will receive 0.9% Sodium Chloride or 5% Dextrose 100ml administered via intravenous infusion over at least 15 minutes on Day 1.
  Other Names: Saline; Placebo
  Arms: Denosumab; Placebo
Drug: Sodium Chloride 0.9% Injection — Patients allocated to the placebo arm and Zoledronic acid arm will receive 0.9% Sodium Chloride 1ml administered via subcutaneous injection on Days 1 and Day 180
  Other Names: Saline; Placebo
  Arms: Placebo; Zoledronic acid

SUMMARY:
The Bone Zone trial is a prospective, multi-centre, double-blind, phase II, randomised controlled trial evaluating the effect of denosumab or zoledronic acid compared to placebo on change in bone mineral density over one year in women aged 50 years or older and men aged 70 years or older requiring admission to intensive care for greater than 24 hours.

450 women aged 50 years or older and men aged 70 years or older, admitted to intensive care for greater than 24 hours will be recruited into the study from participating study centres.

DETAILED DESCRIPTION:
Intensive care patients face health issues that extend beyond their critical illness. A specific area where critical illness may adversely affect the well-being of survivors is increased bone turnover during critical illness, and accelerated bone loss in subsequent years. Critical illness bone loss begins in the first days of critical illness, occurs in both men and women, and is greatest in post-menopausal women. Loss of bone mineral density is significantly greater at both the femur (-2+4.0% vs -0.7+1.1%, p=0.001) and spine (-2.9+4.1% vs -0.2+1.1%, p<0.001) in women in the year after critical illness compared to age-matched controls. One year after critical illness, 80% of women aged 50-years or greater are classified as osteoporotic or osteopaenic, compared to 71% of the approximately 3.7 million Australian women aged 50 year or greater. In the year after ICU admission a decrease in femur BMD of -1.52% (+ 2.85) is reported in men, which is significantly higher than age adjusted population controls (-0.42% + 1.13, diff -1.10% (95% CI -1.71 to -0.49, p<0.001). The annual incidence of first fracture in men aged 70 years and over is similar to the annual incidence of fracture in women aged 50 years and over. In addition, there is a dramatic increase in hip fractures as a proportion of all fracture's males aged 70 years and older in the general population. This population is most likely to suffer the major consequence of accelerated bone loss, fragility fracture, and the associated morbidity, loss of quality of life, and economic cost. Older women who survive critical illness have a significantly higher fragility fracture rate compared to community age-matched controls (Intensive Care Unit 4.33 vs control 2.81 per 100 patient years, adj HR 1.7 (95% CI 1.1-2.5), p=0.02).

Bone antiresorptive therapies are effective at reducing bone loss and decreasing fracture risk in non-critically ill populations. Zoledronic acid and denosumab represent antiresorptive agents with established efficacy in adults, and are potential target interventions able to be delivered during critical illness. Denosumab is a human monoclonal antibody directed against Receptor activator of nuclear factor kappa-Β ligand, a central stimulator of osteoclast activity, and is effective for prevention of fractures and bone loss in osteoporosis and malignancy. Zoledronic acid is a bisphosphonate class agent that binds to bone and suppresses bone resorption by entering osteoclasts and inhibiting the enzyme farnesyl pyrophosphate synthase, resulting in disruption of osteoclast attachment to bone surface. In addition to skeletal effects, there are possible mortality benefits associated with the use of antiresorptive medications in populations with increased bone loss.

There is currently insufficient high-quality evidence to support routine, early use of antiresorptive medications in critically ill adults. The Bone Zone trial is a phase III multi-centre randomised placebo-controlled trial of 450 women aged 50-years or greater and men aged 70-years or greater requiring intensive care admission for more than 2 calendar days, to determine the effect of denosumab or zoledronic acid on the prevention of bone loss in the year after critical illness.

ELIGIBILITY:
Inclusion Criteria:

* Female age ≥ 50 years or male age ≥ 70 years
* Has been in the Intensive Care Unit for 2 or more calendar days and is not expected to be discharged from the Intensive Care Unit on the second day
* Has required Intensive Care Unit level support (i.e. intravenous vasoactive drugs, or invasive mechanical ventilation, or non-invasive ventilation or high flow nasal oxygen at Fraction inspired Oxygen ≥0.4 and/or gas flows ≥40L/m) for a minimum cumulative duration of 6 hours
* Expected to survive the current hospital admission

Exclusion Criteria:

* Cancer related metastatic bone disease or multiple myeloma
* Paget's disease
* Pregnancy
* Current estimated Glomerular Filtration Rate <30ml/min or receiving renal replacement therapy
* Known contraindication to denosumab or zoledronic acid
* Obvious holes in teeth or broken teeth or dental or gum infection
* Known untreated hypoparathyroidism
* Current treatment with anti-fracture agent (bisphosphonate, strontium or teriparatide within previous 2 years, or menopausal hormone therapy or romosozumab within previous 12-months or denosumab within previous 6 months)
* Current fragility fracture of hip, spine, femur or forearm
* Exceeds weight limit for BMD scan at site or unable to undertake Bone Mineral Density for any reason
* International Normalised Ratio > 3.0 or Platelet count < 30 10^9/L

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Annualised change in femoral neck bone mineral density for the year after Intensive Care discharge | 12 months
  Change in femoral neck bone mineral density T-score between baseline and 12 months

SECONDARY OUTCOMES:
Annualised change in lumbar spine bone mineral density for the year after Intensive Care discharge | 12 months
  Change in lumbar spine bone mineral densityT-score between baseline and 12 months
Clinical fragility fracture | 6 and 12 months
  Self-reported incident clinical fractures obtained at follow-up visits. Information on the date, site, and circumstance of the fracture obtained by interview and X-ray report sought and confirmed by medical report.
Vertebral fracture | 12 months
  Incident vertebral fracture obtained during lateral BMD study
Falls | 6 and 12 months
  Self-reported falls incidence and frequency
Hospital readmission | 12 months
  All hospital readmissions within 12 months will be recorded
Mortality | 12 months
  All deaths from enrolment to 12 months will be recorded
Change in quality of life | 0, 6 and 12 months.
  Quality of life will be measured using the European Quality of Life scale using a descriptive system scale from 1 to 5
Bone turnover outcomes (nested sub-study) | Day 0, Day 7, 6 and 12 months
  Change in the bone turnover markers serum collagen type 1 cross-linked c-telopeptide (CTX), and serum type 1 procollagen N-terminal propeptide (P1NP)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Orford, A/Prof, Study Chair — Barwon Health; ANZIC Research Centre; Priya Nair, A/Prof, Study Chair — St Vincent's Health Sydney
Locations (23):
- Australia (21):
  - John Hunter Hospital, Newcastle, New South Wales
  - St Vincent's Health Sydney, Sydney, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Blacktown Hospital, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Wollongong Hospital, Illawarra Shoalhaven Health, Wollongong, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - The Wesley Hospital, Brisbane, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Barwon Health, University Hospital Geelong, Geelong, Victoria
  - Alfred Health, Melbourne, Victoria
  - Western Health - Footscray Hospital, Melbourne, Victoria
  - Western Health - Sunshine Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - St Vincents Hospital Melbourne, Melbourne, Victoria
  - Austin Health, Melbourne, Victoria
  - Eastern Health - Box Hill Hospital, Melbourne, Victoria
  - St John of God Hospital Subiaco, Perth, Western Australia
  - Fiona Stanley Hospital, Perth, Western Australia
  - St John of God Hospital Murdoch, Perth, Western Australia
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Wellington Regional Hospital, Wellington

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of the study, the study management committee will consider requests from researchers who provide a methodologically sound scientific proposal as per the Data Sharing Policy set out in the ANZIC Research Centre Terms of Reference.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: As per the ANZIC Research Centre Data Sharing Policy
Access Criteria: As per the ANZIC Research Centre Data Sharing Policy
URL: https://www.monash.edu/__data/assets/pdf_file/0005/2699411/2023-07-28-ANZIC-RC-Terms-of-Ref.pdf